CLINICAL TRIAL: NCT01929460
Title: A Prospective, Placebo-controlled Trial on the Use of Antibiotics for Pancreatic Cyst Aspiration: a Pilot Study
Brief Title: A Pilot Study on the Use of Prophylactic Antibiotics for EUS-guided Pancreatic Cyst Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2013-08-13; First posted 2013-08-28 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Pancreatic Cysts
MeSH Terms: conditions — Pancreatic Cyst | interventions — Ciprofloxacin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug (Standard group) (Other): Standard group: this group will receive three days of oral antibiotics after their EUS-guided pancreas cyst aspiration.
  Ciprofloxacin 500mg by mouth twice a day for three days.
  Interventions: Drug: Ciprofloxacin
- Intervention group (Placebo Comparator): Intervention group: this group will receive three days of oral PLACEBO after their EUS-guided pancreas cyst aspiration
  Oral Placebo, one cap twice a day for three days.
  Interventions: Other: Placebo (for ciprofloxacin)

INTERVENTIONS:
Drug: Ciprofloxacin — ciprofloxacin oral capsule (one capsule twice a day for 3 days)
  Other Names: Cipro
  Arms: Drug (Standard group)
Other: Placebo (for ciprofloxacin) — oral placebo capsule (one capsule twice a day for 3 days)
  Other Names: sugar pill formulated to mimic oral ciprofloxacin
  Arms: Intervention group

SUMMARY:
Our hypothesis is that a single dose of antibiotics at time of EUS-guided pancreatic cyst aspiration is equally effective to the usual regimen of 3 days of post-procedural antibiotics.

DETAILED DESCRIPTION:
With the increased use of cross sectional imaging, there appears to be an increasing prevalence of pancreatic cysts being incidentally discovered.

A critical step in the workup of pancreas cysts is to determine whether the cyst is mucinous or non-mucinous, through a procedure called endoscopic ultrasound - fine needle aspiration (EUS-FNA).

Current guidelines suggest the use of antibiotics in cyst aspiration, usually 3 days after the procedure. However, these recommendations are based on limited data from over 15 years ago. More recent retrospective observations suggest equivalent safety when little, or even no antibiotics are given.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18-90 who present for an EUS / pancreas cyst evaluation

Exclusion Criteria:

* Patients outside the age range
* Patient-related factors (unable to provide consent, unable to understand English, allergic to cipro)
* High-risk patients for infective endocarditis
* Bacterial infection or use of antibiotics within 6 weeks of EUS
* Pancreatitis within the past 6 months
* Underlying immunosuppression (for example, uncontrolled diabetes - such as hemoglobin A1c above 7 or glucose > 180; renal failure; cirrhosis; pre-existing malignancy especially hematologic malignancy such as leukemia / lymphoma / multiple myeloma; HIV/AIDS)
* Currently taking immunosuppressive medications (for conditions such as rheumatoid arthritis, inflammatory bowel disease, organ transplant)
* Radiographic or endosonographic evidence of cyst cavity debris / necrotic debris
* Severe systemic disease (for example, NYHA class III or IV heart failure, oxygen-dependent COPD)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Kwok, MD, Principal Investigator — Principal Investigator
Locations (1):
- Kaiser Permanente, Los Angeles Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Jacobson BC, Baron TH, Adler DG, Davila RE, Egan J, Hirota WK, Leighton JA, Qureshi W, Rajan E, Zuckerman MJ, Fanelli R, Wheeler-Harbaugh J, Faigel DO; American Society for Gastrointestinal Endoscopy. ASGE guideline: The role of endoscopy in the diagnosis and the management of cystic lesions and inflammatory fluid collections of the pancreas. Gastrointest Endosc. 2005 Mar;61(3):363-70. doi: 10.1016/s0016-5107(04)02779-8. No abstract available. PMID 15758904
- [Background] Lee LS, Saltzman JR, Bounds BC, Poneros JM, Brugge WR, Thompson CC. EUS-guided fine needle aspiration of pancreatic cysts: a retrospective analysis of complications and their predictors. Clin Gastroenterol Hepatol. 2005 Mar;3(3):231-6. doi: 10.1016/s1542-3565(04)00618-4. PMID 15765442

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciprofloxacin (Standard Group): Standard group: this group will receive three days of oral antibiotics after their Endoscopic Ultrasound (EUS)-guided pancreas cyst aspiration.
  Ciprofloxacin 500mg by mouth twice a day for three days.
  Ciprofloxacin
- Placebo (Intervention Group): Intervention group: this group will receive three days of oral PLACEBO after their Endoscopic Ultrasound (EUS)-guided pancreas cyst aspiration
  Oral Placebo, one cap twice a day for three days.
  Placebo (for ciprofloxacin)
Period: Overall Study
Arm/Group | Ciprofloxacin (Standard Group) | Placebo (Intervention Group)
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ciprofloxacin (Standard Group): Standard group: this group will receive three days of oral antibiotics after their EUS-guided pancreas cyst aspiration.
  Ciprofloxacin 500mg by mouth twice a day for three days.
  Ciprofloxacin
- Placebo (Intervention Group): Intervention group: this group will receive three days of oral PLACEBO after their EUS-guided pancreas cyst aspiration
  Oral Placebo, one cap twice a day for three days.
  Placebo (for ciprofloxacin)
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin (Standard Group) | Placebo (Intervention Group) | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Full Range); unit: years] | 68 [40 to 85] | 68.5 [50 to 82] | 68.3 [40 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
Number of fine needle aspiration (FNA) passes [Mean (Full Range); unit: passes] | 1.46 [1 to 3] | 1.38 [1 to 3] | 1.42 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pancreas Cyst Infection After EUS-guided Pancreatic Cyst Aspiration
Description: first time point (number of patients with pancreas cyst infection after EUS-guided pancreatic cyst aspiration)
Time Frame: At 2 weeks after procedure
Measure: Number; unit: participants
Arm/Group | Ciprofloxacin (Standard Group) | Placebo (Intervention Group)
Number analyzed (Participants) | 13 | 13
participants | 0 | 0

2. Primary Outcome: Number of Patients With Pancreas Cyst Infection After EUS-guided Pancreatic Cyst Aspiration
Description: second time point (number of patients with pancreas cyst infection after EUS-guided pancreatic cyst aspiration)
Time Frame: At 4 weeks after procedure
Measure: Number; unit: participants
Arm/Group | Ciprofloxacin (Standard Group) | Placebo (Intervention Group)
Number analyzed (Participants) | 13 | 13
participants | 0 | 0

3. Primary Outcome: Number of Patients With Pancreas Cyst Infection After EUS-guided Pancreatic Cyst Aspiration
Description: third and final time point (number of patients with pancreas cyst infection after EUS-guided pancreatic cyst aspiration)
Time Frame: At 6 weeks after procedure
Measure: Number; unit: participants
Arm/Group | Ciprofloxacin (Standard Group) | Placebo (Intervention Group)
Number analyzed (Participants) | 13 | 13
participants | 0 | 0

4. Secondary Outcome: Adverse Drug Reactions
Description: Number of participants with adverse drug reactions
Time Frame: six weeks
Measure: Number; unit: participants
Arm/Group | Ciprofloxacin (Standard Group) | Placebo (Intervention Group)
Number analyzed (Participants) | 13 | 13
participants | 0 | 0

5. Secondary Outcome: Procedure-related Complications
Description: Number of patients with procedure-related complications
Time Frame: six weeks after procedure
Measure: Number; unit: participants
Arm/Group | Ciprofloxacin (Standard Group) | Placebo (Intervention Group)
Number analyzed (Participants) | 13 | 13
participants | 0 | 5

6. Secondary Outcome: Mean Cyst Fluid Carcinoembryonic Antigen (CEA)
Description: Mean cyst fluid carcinoembryonic antigen (CEA) for classification of mucinous cystic lesions
Time Frame: six weeks
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Ciprofloxacin (Standard Group) | Placebo (Intervention Group)
Number analyzed (Participants) | 13 | 13
ng/mL | 214.1 [0.2 to 1982] | 2466.2 [0.2 to 24056]

7. Secondary Outcome: Mean Cyst Fluid Amylase
Description: Mean cyst fluid amylase for classification of mucinous cystic lesions
Time Frame: six weeks
Measure: Mean (Full Range); unit: Units/L
Arm/Group | Ciprofloxacin (Standard Group) | Placebo (Intervention Group)
Number analyzed (Participants) | 13 | 13
Units/L | 3729 [30 to 7200] | 1944.5 [28 to 7200]

8. Secondary Outcome: Median Cyst Fluid Carcinoembryonic Antigen (CEA)
Description: Median cyst fluid carcinoembryonic antigen (CEA) for classification of mucinous cystic lesions
Time Frame: six weeks
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Ciprofloxacin (Standard Group) | Placebo (Intervention Group)
Number analyzed (Participants) | 13 | 13
ng/mL | 15 [3.4 to 74.5] | 24.9 [0.35 to 248.5]

9. Secondary Outcome: Median Cyst Fluid Amylase
Description: Median cyst fluid amylase for classification of mucinous cystic lesions
Time Frame: six weeks
Measure: Median (Inter-Quartile Range); unit: Units/L
Arm/Group | Ciprofloxacin (Standard Group) | Placebo (Intervention Group)
Number analyzed (Participants) | 13 | 13
Units/L | 4006.5 [167.5 to 7200] | 239 [144 to 2930]

ADVERSE EVENTS:
Time Frame: Adverse events were prospectively monitored during the study period (1/1/2014-12/31/2014) at 2, 4, 6 weeks post procedure, or if the patient contacted the on-call research staff at any time after hours.
Groups:
- Drug (Standard Group): Standard group: this group will receive three days of oral antibiotics after their EUS-guided pancreas cyst aspiration.
  Ciprofloxacin 500mg by mouth twice a day for three days.
  Ciprofloxacin
- Intervention Group: Intervention group: this group will receive three days of oral PLACEBO after their EUS-guided pancreas cyst aspiration
  Oral Placebo, one cap twice a day for three days.
  Placebo (for ciprofloxacin)
Arm/Group | Drug (Standard Group) | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/13
Other Adverse Events (participants affected / at risk) | 0/13 | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug (Standard Group) (N=13) | Intervention Group (N=13)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — one patient in the placebo arm was admitted for post-procedure pancreatitis. Recovered without incident.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug (Standard Group) (N=13) | Intervention Group (N=13)
pain (Gastrointestinal disorders) | 0 (0) | 4 (4) — 2 cases deemed unrelated to the procedure (1, nephrolithiasis; 1, chronic abdominal pain). 1 case deemed probably unrelated 1 case deemed possibly related but resolved uneventfully with conservative measures only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes